CLINICAL TRIAL: NCT06781411
Title: Unity Cures Future (UCF) Biobank for Translational & Biomedical Research At UCF College of Medicine and Burnett School of Biomedical Sciences with Identifiable Human Tissue.
Brief Title: Unity Cures Future (UCF) Biobank
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00007256
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Tissue Banking
Keywords: tissue; donate; surgery; biobank

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Donated Human Tissue: This Project will receive discarded human tissue from consented participants. For the purposes of this project, human tissue is defined as any bodily material collected from a human person, including bone marrow, skin, tumors, etc., through a clinical procedure. The clinical procedure will done not be done solely for the purpose of this Project. Participants (donors) will prospectively provide informed consent, complete an online case report form, and donate the unwanted human tissue that results from their surgery/procedure.

SUMMARY:
Research scientists of the University of Central Florida College of Medicine (COM) and Burnett School of Biomedical Sciences (BSBS) conduct laboratory studies in biomedical and translational medical research for the purpose of understanding human disease and developing innovative methods for diagnosing, measuring, or treating disease or disease symptoms. The key research divisions are cancer, cardiovascular, immunity and pathogenesis, neuroscience, and molecular microbiology.

DETAILED DESCRIPTION:
The goal of this human tissue repository protocol is to aggregate resources and streamline the acquisition of human tissue. It is optimal for the advancement of biomedical and translational medical research that the human tissue be received under one protocol by the College of Medicine's the Clinical & Aerospace Health Research team and transferred to the COM/BSBS research scientists for laboratory testing.

This aggregation of efforts and resources through a human tissue repository protocol allows for:

1. Improvements in biomedical and translational medical research by availability of viable human tissues.
2. Reduced recruitment and enrollment burden on the Clinical & Aerospace Health Research team and the participants via pooled recruitment. Further, participants will only need to provide one informed consent. Received human tissue may be used for multiple protocols.
3. Improved data for analysis as participants will complete an online case report form containing basic demographic data; planned location and date of upcoming surgery or procedure; diagnosis; name of surgeon/doctor for the planned surgery or procedure; type of surgery or procedure; medical data; medical history; and surgery history.

ELIGIBILITY:
Inclusion Criteria:

1. be able to read and understand English
2. scheduled for a surgery or procedure that will result in the removal of human tissue.

Exclusion Criteria:

1. Pregnant
2. unable to provide an informed consent
3. unable to understand or read in English
4. minors (ages under 18)
5. prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will donate unwanted human tissue as a result of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2075-11-06 (Estimated); Study Completion 2075-11-06 (Estimated)

PRIMARY OUTCOMES:
Receipt of donated human tissue for research | 50 years
  The key research divisions are cancer, cardiovascular, immunity and pathogenesis, neuroscience, and molecular microbiology. Frequently, these studies require human tissue for testing of assays and devices.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States